CLINICAL TRIAL: NCT04963712
Title: A Prospective Single-arm Cohort Study Evaluating the Safety and Efficacy of Thymalfasin (Zadaxin®) in the Treatment of HIV-positive Patients With Immune Reconstitution Disorders
Brief Title: Zadaxin and HIV-positive Patients With Immune Reconstitution Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, Professor, Shanghai Public Health Clinical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zadaxin-HIV
Record Dates: First submitted 2021-07-07; First posted 2021-07-15 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Thymalfasin

STUDY DESIGN:
Intervention Model Description: All participants eligible for study received the same open label drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zadaxin-HIV(n=20) (Experimental): Study participants will be given Zadaxin (1.6 mg subcutaneous injection, once a day) in the first 2 weeks, and changed frequency (1.6 mg subcutaneous injection, twice a week) in the successive 22 weeks.
  Interventions: Drug: Zadaxin

INTERVENTIONS:
Drug: Zadaxin — 1.6 mg subcutaneous injection, once a day in the first 2 weeks, and 1.6 mg subcutaneous injection, twice a week in the successive 22 weeks.
  Other Names: Thymosin α1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Zadaxin® in the treatment of HIV-positive patients with immune reconstitution disorders. Researchers previously used Zadaxin® (Thymosin α-1, Tα1) as an immune adjuvant for people infected with HIV-1 and found that Tα1 and Interferon-α (IFN-α) have a synergistic effect in immune enhancement. In addition, studies have found that the triple combination of Tα1, IFN-α and Zidovudine has better tolerability, safety and efficacy. After treatment, patients have lower HIV RNA and more stable high CD4+ T cell counts. In addition, extensive studies on the administration of Tα1 in thymectomized mice have demonstrated its ability to promote immune reconstitution. The researchers hypothesized that Zadaxin® has a better therapeutic effect on HIV-positive patients with immune reconstitution disorders, can increase the CD4+T cell count, reduce the viral load, and has better safety.

DETAILED DESCRIPTION:
All patients received Zadaxin (1.6 mg subcutaneous injection, once a day) in the first 2 weeks, and changed frequency (1.6 mg subcutaneous injection, twice a week) in the successive 22 weeks. It is still recommended to continue treatment until the end of the study. All subjects were given HAART treatment throughout. In 4th week, 8th week, 12th week and 24th week, perform 4 follow-up and record the changes in CD4+ T cell count and proportion, CD8+ T cell count and proportion, proportions of T cell subsets, PBMC sjTREC, proportions of exhauseted T cell expressed PD-1 and Tim-3, and HIV viral load. During the process, safety assessment is performed, including adverse events, electrocardiogram and a series of laboratory tests (blood routine, liver and kidney function, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old;
* HIV serology is positive;
* Volunteer to participate;
* CD4+T cell count >100 and <350 cells/mm3;
* People who have received HAART treatment and the viral load is undetected for at least 2 years, but have immune reconstitution disorder;
* Without active opportunistic infection;

Exclusion Criteria:

* History of allergy or contraindications to Zadaxin;
* Skin basal cell carcinoma, cervical carcinoma in situ or other concurrent tumors other than Kaposi's sarcoma;
* The expected survival time is less than 1 year;
* Women of childbearing age have a positive pregnancy test;
* Major heart disease or central nervous system disease or other nervous system abnormalities;
* ACTG-AIDS dementia syndrome staging score> 0.5;
* Organ transplantation;
* Received chemotherapy and radiotherapy for malignant tumors within 6 months;
* Known immunomodulators (such as systemic steroids, interferons, interleukins) or other immunotherapy within 30 days before the start of the study;
* Blood transfusion within 30 days before the start of the study;
* Have a history of iritis, endophthalmitis, scleritis or retinitis;
* Within 30 days before the screening assessment, accept any experimental treatment for HIV-positive patients with or without symptoms of infection;
* Drug abuse;
* The doctor's decision is that participation in the trial is not in the patient's best interests, or any situation that does not allow safe compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Change in CD4+T cell counts | Measured on week 24
  Peripheral blood
Change in CD4/CD8 ratio | Measured on week 24
  Peripheral blood

SECONDARY OUTCOMES:
Change in CD4+T cell count and proportion | Measured on week 0, 4, 8, 12, 24
  Peripheral blood
Change in CD8+T cell count and proportion | Measured on week 0, 4, 8, 12, 24
  Peripheral blood
Change in proportions of T cell subsets | Measured on week 0, 4, 8, 12, 24
  Peripheral blood mononuclear cell
Change in proportions of immune exhausted T cells expressed PD-1 and TIM-3 | Measured on week 0, 4, 8, 12, 24
  Peripheral blood mononuclear cell
Change in PBMC sjTREC | Measured on week 0, 4, 8, 12, 24
  Peripheral blood mononuclear cell
Change in HIV-1 RNA | Measured on week 0, 4, 8, 12, 24
  Plasma

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Ph.D, Study Director — Shanghai Public Health Clinical Center
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen C, Wang J, Xun J, Zhang X, Liu L, Song Z, Zhang R, Chen J, Lu H. Role of thymosin alpha1 in restoring immune response in immunological nonresponders living with HIV. BMC Infect Dis. 2024 Jan 17;24(1):97. doi: 10.1186/s12879-024-08985-y. PMID 38233816